CLINICAL TRIAL: NCT05500846
Title: Targeted Cryoablation of Prostate Cancer Lesions: An Investigator-initiated Trial
Acronym: PROCRY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Osamu Ukimura (Other)
Responsible Party: Sponsor-Investigator, Osamu Ukimura, Professor, Department of Urology, Kyoto Prefectural University of Medicine
Organization: Kyoto Prefectural University of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTREC-URO-181202; jRCT2052210088 (Other: Japan Registry of Clincal Trials)
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Localized Prostate Cancer; CISca, Clinically Insignificant Prostate Cancer; CSCa, Clinically Significant Prostate Cancer; Focal Therapy; Treatment of partial prostate; Cryotherapy; Cryosurgery; Targeted Cryoablation; Ultrasound guided surgery; Targeted Prostate Biopsy; MRI, Magnetic Resonance Imaging; PSA, Prostate Specific Antigen; QOL, Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms; Salivary Gland Adenoma, Pleomorphic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cryoablation Arm (Experimental): Minimally invasively trans-perineal puncture of both cryo-needles and temperature-needles will be placed under real-time image guidance to the targeted area of cancer lesion or temperature-monitoring sites, respectively. The targeted tissue surrounding the tip of cryo-needles will be freeze down to targeted temperature for killing the cancer cells, and other non-treated area will be left in the prostate for aiming of maintain QOL (quality-of-life). The Minimally invasive cryoablation surgery will be performed under general anesthesia within one and half hour for aiming to be provided total 50 patients. (The used device for this arm has been clinically approved for cryoablation of renal cancer in Japan.)
  Interventions: Device: The Visual Ice Cryoablation System

INTERVENTIONS:
Device: The Visual Ice Cryoablation System — Currently, the standard surgical treatment option for localized prostate cancer is total prostatectomy, which removes the entire prostate organ. However, total prostatectomy is invasive and postoperative urinary incontinence, sexual dysfunction and local recurrence remain clinical challenges even with the introduction of robotic assistance techniques. Cryotherapy has been approved as one of the other surgical treatment options for localized prostate cancer in the USA and Europe, but not in Japan. This clinical trial aims to expand the indication of cryotherapy equipment, which has already been approved for insurance for renal cancer, to prostate cancer in Japan. In this clinical trial, Focal Therapy will be performed by targeting a single localized prostate cancer lesion visualized by MRI. By targeting cancer lesions in a minimally invasive manner, we aim to achieve both control of cancer lesions and maintenance of quality of life.
  Other Names: Targeted focal cryoablation of localized prostate cancer

SUMMARY:
This clinical trial is to provide a minimally invasive treatment option in which the targeted prostate cancer tissue is killed by cryoablation at extremely low temperatures only in the specific area of cancer "that should be treated for saving of life"; while, leaving a portion of the normal prostate tissue that is not cancerous. It is a treatment, named by "focal therapy" for "clinically localized prostate cancer". As this new treatment is aiming to treat only specific prostatic area of cancer, it is different from the invasive conventional treatment to remove the entire prostate gland. The goal is to achieve both to control of known cancer by treating only the cancerous area and to maintain of QOL (Quality-of-life) by leaving of the other normal prostate tissue and its surrounding organs intact resulting in prevention of urinary-leakage and sexual-dysfunction as the complications.

DETAILED DESCRIPTION:
This trial will to provide an ultrasound-guided targeted cryoablation of known cancer lesions in patients diagnosed with clinically localized prostate cancer, and this trial will assess effectiveness for up to post-operative 6 months and safety for up to postoperative 12 months. This trial will assess patient quality of life (QOL) as well.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have a PI-RADS category 3 or 4 lesion on MRI image at enrollment and who have a single lesion with a Gleason score 7 or 8 on histopathology of the prostate needle biopsy at enrollment; or, patients who have a PI-RADS category 4 or 5 lesion on MRI image at enrollment and who have a single lesion with a Gleason score 6 or 7 on histopathology of the prostate needle biopsy at enrollment
2. Patients with prostate cancer that is clinical stage T2c or lower (T1a-T2cN0M0) according to the TNM Classification as determined during enrollment
3. Patients between the ages of 20 and 85 when providing consent to participate in this trial
4. Patients from whom consent is obtained prior to enrollment in this trial

Exclusion Criteria:

1. Patients to have a lesion identified as PI-RADS category 4 or 5 on MRI images at enrollment and who have a single lesion with a diameter of less than 10 mm and Gleason score of 6 on the histopathology of the prostate needle biopsy at enrollment (the lesion is referred to as "non-target lesions") (the diameter of the lesion is defined as the longer one of the lesion diameter identified on MRI images at enrollment or the tumor length as measured on histopathology of prostate needle biopsy)
2. Patients to have 4 or more non-target lesions (non-target lesions are defined as the lesions defined in exclusion criterion 1, or lesions with PI-RADS category 3 on MRI image at enrollment and Gleason score 6 on biopsy at enrollment)
3. Patients to have a lesion with PI-RADS category 5 on MRI image at enrollment and Gleason score 8 on histopathology of prostate needle biopsy at enrollment (the lesion is referred "excluded lesions")
4. Patients with a serum prostate-specific antigen (PSA) level over 20 ng/ml during enrollment
5. Patients in whom the distance from the target prostate cancer lesion to an external urinary sphincter is 5 mm or less on MRI images (coronal or sagittal) obtained during enrollment
6. Patients who have undergone surgery, drug therapy, or radiation therapy for prostate cancer prior to enrollment
7. Patients who have received an antiandrogen for benign prostatic hyperplasia prior to enrollment
8. Patients using absorbent pads or adult diapers due to urge incontinence
9. Patients with active multiple cancers
10. Patients for whom MRI scans are contraindicated
11. Patients in whom transrectal ultrasound cannot be performed for some reason, such as a constricted rectum
12. Patients with a prothrombin time<50% or platelet count<60,000/mm3 during enrollment
13. Patients deemed to be ineligible by an investigator

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Because the prostate is an organ that only men have.
Enrollment: 51 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disappearance of cancer at 6 month after cryosurgery evaluated by combination of the responses in PSA, MRI, and Prostate biopsy | 6 months after the cryosurgery
  Achievement of all endpoints in the three clinical parameters including 1) reduction of serum PSA value, 2) reduction of PI-RADS category for MRI-visible lesion, and 3) histological disappearance of cancer by prostate biopsy
  1. A 50% or greater reduction from the preoperative serum PSA level at postoperative 3 or 6 months
  2. A reduction of PI-RADS category of the targeted prostate cancer lesion down to 3 or lower at MRI images at postoperative 6 months
  3. No cancer tissue in histopathological examination from the targeted prostate cancer lesion via a needle biopsy of the prostate performed at postoperative 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Ukimura, M.D., Ph.D., Principal Investigator — Department of Urology, University Hospital, Kyoto Prefectural University of Medicine; Toshiko Ito-Ihara, M.D., Ph.D., Study Chair — The Clinical and Translational Research Center , University Hospital, Kyoto Prefectural University of Medicine (CTREC)
Locations (2):
- Japan (2):
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Kyoto Miniren Chuo Hospital, Kyoto

IPD SHARING:
Plan to Share IPD: No